CLINICAL TRIAL: NCT06369181
Title: Neuroendocrine Transformation in RB1 and TP53 Inactivated Non-small Cell Lung Cancer Patients: a Multi-center Prospective Observational Study
Brief Title: Neuroendocrine Transformation in RB1/TP53 Inactivated NSCLC
Status: Recruiting | Type: Observational
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhengfei Zhu, Chief physician, Department of Radiation Oncology, Fudan University
Other Study IDs: NET 2020
Record Dates: First submitted 2024-04-12; First posted 2024-04-16 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Neuroendocrine Carcinoma; Non-small Cell Lung Cancer; Histology Transformation
Keywords: neuroendocrine transformation; small cell lung cancer transformation; TP53; RB1; histology transformation; non-small cell lung cancer
MeSH Terms: conditions — Carcinoma, Neuroendocrine; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Histology transformation from non-small cell lung cancer (NSCLC) to neuroendocrine carcinomas (NEC), especially from epidermal growth factor receptor (EGFR) mutant lung adenocarcinoma (LADC) to small cell lung cancer (SCLC), is widely recognized as a rare mechanism for NSCLC to confer tyrosine kinase inhibitors (TKIs) resistance. The probability of its occurrence is about 3-14% in NSCLC patients who are resistant to TKI treatment. In addition to EGFR mutations, NSCLC patients carrying ALK/ROS1 mutations and receiving corresponding TKI treatment may also experience NEC transformation(NET).

In a previous study [Pubmed ID: 35609408], the investigators demonstrated that NET also develops in NSCLCs without TKI targets or treatments. This phenomenon could be under-recognized, because re-biopsy was less frequently performed in these patients. The investigators had also shown that p53/Rb inactivation might correlated with NET and should be considered for NET risk prediction. In another retrospective studies, it was found that NSCLC patients with RB1/TP53 dual inactivation mutations had a significantly higher probability of NEC pathological transformation than those without RB1/TP53 inactivation mutations (43 times higher than those without mutations). Therefore, the subgroup of NSCLC patients with tumor suppressor gene RB1/TP53 dual inactivation might have elevated risk for NET.

In this study, the investigators proposed to prospectively follow up NSCLC patients with dual RB1/TP53 inactivation (approximately 5% of the total NSCLC). Through prospective and systematic collection of baseline pathological information, clinical treatment process, and imaging data, and as much as possible, repeat pathological biopsies will be performed during disease progression.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old;
2. ECOG function status score 0-2 points;
3. Pathological diagnosis of stage III-IV non neuroendocrine non-small cell lung cancer;
4. RB1/TP53 gene/protein testing (IHC, NGS, or other techniques are acceptable) has been completed and confirmed to be dual inactivation of RB1/TP53;
5. For patients with baseline pathology of adenocarcinoma, complete driver gene testing (including at least EGFR and ALK);
6. The patient undergoes at least one systemic treatment (chemotherapy, targeted drug therapy, immunotherapy, etc.) and receives regular follow-up;
7. After discovering disease progression during the follow-up process, the patient will undergo further pathological biopsy of the progressing lesion after evaluation by the sub center PI;
8. According to the researcher's assessment, the patient currently does not require palliative radiation therapy in any area;
9. If the subject undergoes surgery, they must fully recover from the toxicity and complications of the surgical intervention before starting treatment;
10. The subjects need to agree to provide corresponding peripheral blood and biopsy tissue samples before and during the follow-up treatment in accordance with the clinical trial protocol requirements;
11. Men/women of childbearing age agree to use contraception during the trial period (surgical ligation or oral contraception/intrauterine device+condom contraception);
12. Life expectancy ≥ 3 months;
13. Patients must have the ability to understand and voluntarily sign informed consent forms.

Exclusion Criteria:

1. Baseline pathological examination reveals neuroendocrine components (including any percentage of small cell carcinoma, large cell carcinoma, differentiated neuroendocrine carcinoma, etc);
2. Unable to perform RB1/TP53 testing ;
3. Patients with baseline pathology of adenocarcinoma and inability to perform driver gene testing (including at least EGFR, ALK);
4. Symptomatic interstitial lung disease or active infection/non infectious pneumonia;
5. History of other malignant tumors;
6. Physical examination or clinical trial findings that researchers believe may interfere with the results or increase the risk of treatment complications for patients, or other uncontrollable diseases
7. Breastfeeding or pregnant women;
8. Congenital or acquired immunodeficiency diseases, including human immunodeficiency virus (HIV), or a history of organ transplantation or allogeneic stem cell transplantation;
9. Patients who require long-term treatment with cortisol or immunosuppressants;
10. Patients with mental illnesses, substance abuse, or social issues that affect compliance will not be included in the group after being reviewed by a doctor
11. Individuals who receive other long-term medication treatments and have been assessed by a doctor as potentially affecting disease progression.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: stage III-IV non-small cell lung cancer with baseline TP53 and RB1 inactivations.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
neuroendocrine transformation rate | 10 years after enrollment
  Number of patients developed neuroendocrine transformation and its proportion in the entire progressed cohort

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Background] Chu X, Xu Y, Li Y, Zhou Y, Chu L, Yang X, Ni J, Li Y, Guo T, Zheng Z, Zheng Q, Yao Q, Li Y, Zhou X, Zhu Z. Neuroendocrine transformation from EGFR/ALK-wild type or TKI-naive non-small cell lung cancer: An under-recognized phenomenon. Lung Cancer. 2022 Jul;169:22-30. doi: 10.1016/j.lungcan.2022.05.002. Epub 2022 May 17. PMID 35609408